CLINICAL TRIAL: NCT01455233
Title: Phase IV Study: A Prospective Two-Site Study to Evaluate the Safety and Tolerance of Besivance Versus Vigamox Prophylactically Pre and Post Operatively in Subjects Undergoing Routine Cataract Surgery
Brief Title: 2-Site Safety Study of Besivance Versus Vigamox Prophylactically in Routine Cataract Surgery
Acronym: STB-01
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ophthalmology Consultants, Ltd. (Other)
Collaborators: Ophthalmology Associates, St Louis (Other); Bausch & Lomb Incorporated (Industry)
Responsible Party: Principal Investigator, Joseph Gira, M.D., Principal Investigator, Ophthalmology Consultants, Ltd.
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: STB-01
Record Dates: First submitted 2011-10-17; First posted 2011-10-19 (Estimated); Last update posted 2011-10-19 (Estimated); Status verified 2010-12

CONDITIONS: Corneal Health; Cataract Surgery
Keywords: cornea; ocular antibiotic; cataract surgery
MeSH Terms: conditions — Corneal Diseases | interventions — besifloxacin; Moxifloxacin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- besivance (Active Comparator): ocular antibiotic
  Interventions: Drug: vigamox
- vigamox (Active Comparator): ocular antibiotic
  Interventions: Drug: besivance

INTERVENTIONS:
Drug: besivance — topical ocular antibiotic, 1 drop in study eye QID starting 3 days prior and for 7 days following cataract surgery
  Other Names: besifloxacin ophthalmic suspension 0.6%
  Arms: vigamox
Drug: vigamox — topical ocular antibiotic, 1 drop in study eye QID for 3 days prior and for 7 days following cataract surgery
  Other Names: moxifloxacin hydrochloride ophthalmic solution 0.5%
  Arms: besivance

SUMMARY:
The purpose of this study is to demonstrate that Besivance is equal to Vigamox in safety and tolerance when used prophylactically in subjects undergoing routine cataract surgery.

DETAILED DESCRIPTION:
Subjects will be assigned to receive either Besivance or Vigamox (1:1) to be administered as 1 drop in the study eye 4 times daily starting 3 days prior to cataract surgery and continuing for 7 days post-operatively.

Sixty subjects (30 from Ophthalmology Consultants and 30 from Ophthalmology Associates) of any race and either sex, requiring cataract extraction with planned implantation of a posterior chamber intraocular lens.

ELIGIBILITY:
Inclusion Criteria:

* Men or woen of any race, 18 years or older who have a cataract, and are planning to undergo cataract extraction by phacoemulsification with the implantation of a posterior chamber intraocular lens
* Study eye of patients who, in the opinion of the investigator, will experience improvement in visual acuity following surgery
* Patients who are able to understand and sign an informed consent form that has been approved by an IRB

Exclusion Criteria:

* Planned multiple procedures during cataract/IOL implantation surgery. Note: A planned limbal relaxing incision may be performed for the correction of astigmatism
* Use of topical ocular or systemic antibiotics within 14 days prior to surgery and through study exit
* History of or Fuch's Corneal Endothelial Dystrophy
* Any ocular inflammation (aqueous cells or flare greater than Grade 0) or ocular pain in the study eye that is present during the baseline visit.
* Recent (within 6 months) ocular trama to the operative eye (this includes intraocular surgery)
* A history of chronic or recurrent inflammatory eye disease (eg, iritis, scleritis, uveitis, iridocyclitis, rubeosis iridis) in the operative eye
* Currently diagnosed uncontrolled glaucoma in the operative eye
* Congenital ocular anomaly (eg, aniridia, congenital cataract) in the operative eye
* A visually nonfunctional fellow eye defined as a best corrected visual acuity </= 35 ETDRS letters (20/200 Snellen equivalent) or worse
* Participation in any other investigational drug or device study within 30 days before cataract surgery
* Known or suspected allergy or hypersensitivity to any component of either test article
* Women of childbearing potential (those who are not surgically sterilized or post menopausal) may not participate in the study if any of the following conditions exist:

  1. they are breast feeding
  2. they have a positive urine pregnancy test at screening
  3. they are not willing to undergo a urine pregnancy test upon entering or exiting the study
  4. they intend to become pregnant during the duration of the study; or,
  5. they do not agree to use adequate birth control methods for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
corneal health | through day 28 post op
  Endothelial Cell Count (day 7, day 28) Pachymetry (day 7, day 28) Corneal Fluorescein Staining (day 7, day 28) Biomicroscopy (day 1, day 7, day 28)

SECONDARY OUTCOMES:
subject tolerance | day - 3 through day 28
  reported adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ranjan Maholtra, MD, Principal Investigator — Ophthalmology Associates; Joseph Gira, MD, Principal Investigator — Ophthalmology Consultants
Locations (2):
- United States (2):
  - Ophthalmology Associates, St Louis, Missouri
  - Ophthalmology Consultants, Ltd, St Louis, Missouri